CLINICAL TRIAL: NCT03580889
Title: Comparison of Atropine Versus Glycopyrrolate in Preventing Spinal Anesthesia Induced Hypotension in Adult Patient Undergoing Major Lower Limb Orthopedic Surgeries
Brief Title: Atropine Versus Glycopyrrolate in Preventing Spinal Anesthesia Induced Hypotension in Lower Limb Surgeries
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Raju Thapamagar, Principal investigator, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRC/1087/017
Record Dates: First submitted 2018-06-17; First posted 2018-07-10 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Lower Extremity Fracture
MeSH Terms: interventions — Atropine; Glycopyrrolate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Atropine sulphate (Active Comparator): Atropine 5 mcg/kg diluted in normal saline to total volume of 2 ml is given intravenous 1 minute after giving intrathecal Bupivacaine 0.5% (Heavy) and patients vitals such as blood pressure, heart rate, SPO2 are monitored every 1 minute for 5 minutes ,then every 5 minutes for 30 minutes then every 10 minutes till end of surgery. Patient shifted to PACU where above vitals are monitored for 2 hrs then shifted to ward. Mean while any adverse outcomes such as nausea, vomiting, sweating, dry mouth is noted and treated accordingly
  Interventions: Drug: Atropine
- Glycopyrrolate (Active Comparator): Glycopyrrolate 2.5 mcg / kg diluted in normal saline to total volume of 2 ml is given intravenous 1 minute after giving intrathecal Bupivacaine 0.5% (Heavy) and patients vitals such as blold pressure, heart rate, SPO2 are monitored every 1 minute for 5 minutes ,then every 5 minutes for 30 minutes then every 10 minutes till end of surgery. Patient shifted to PACU where above vitals are monitored for 2 hrs then shifted to ward. Mean while any adverse outcomes such as nausea, vomiting, sweating, dry mouth is noted and treated accordingly.
  Interventions: Drug: Glycopyrrolate
- Normal Saline (Active Comparator): Normal saline 2 ml is given intravenous 1 minute after giving intrathecal Bupivacaine 0.5% (Heavy) and patients vitals such as blold pressure, heart rate, SPO2 are monitored every 1 minute for 5 minutes ,then every 5 minutes for 30 minutes then every 10 minutes till end of surgery. Patient shifted to PACU where above vitals are monitored for 2 hrs then shifted to ward. Mean while any adverse outcomes such as nausea, vomiting, sweating, dry mouth is noted and treated accordingly.
  Interventions: Drug: Normal Saline Flush, 0.9% Injectable Solution

INTERVENTIONS:
Drug: Atropine — Comparison between atropine, glycopyrrolate and Normal Saline
  Arms: Atropine sulphate
Drug: Glycopyrrolate — Comparison between glycopyrrolate, atropine and Normal saline
  Arms: Glycopyrrolate
Drug: Normal Saline Flush, 0.9% Injectable Solution — Comparison between Normal saline, atropine and glycopyrrolate
  Other Names: Normal Saline
  Arms: Normal Saline

SUMMARY:
A study to compare between intravenous atropine and glycopyrrolate in preventing spinal anesthesia induced hypotension in patients undergoing major lower limb orthopedic surgeries. Hypotension is the most common complication in spinal anesthesia that can be life threatening. If this can be prevented patients comfort can be increased and satisfaction as well.

ELIGIBILITY:
Inclusion Criteria:

* ASA PS I and II,
* age 16 to 65,
* undergoing lower limb major orthopedic surgery,
* willing to participate

Exclusion Criteria:

* Contra indication to spinal anesthesia,
* patient refusal,
* ASA PS >III,
* cardiac diseases,
* hypertension >160/ 100,
* arrhythmias,
* Acute coronary syndrome,
* patients taking beta-blockers,
* hepatic and pulmonary diseases

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Blood pressure from base line will be measured and hypotension will be described and treated as in description section | From anesthesia to 2 hrs after completion of surgery
  Systolic arterial pressure <90 mm of hg or 20% decrease from base line or decrease in blood pressure 30 mm Hg or more from base line will be considered hypotension.
  Hypotension along with tachycardia (as described below) will be treated with phenylephrine 100 mcg and hypotension alone will be treated with mephentermine 6 mg bolus
Heart rate will be monitored and treated accordingly | Iv atropine or glycopyrrolate to 2 hrs after completion of surgery
  Heart rate > 100 Bpm or more or more than 20% from base line will be described as tachycardia. Heart rate less than 50 bpm or less than 20% from baseline will be described as bradycardia

SECONDARY OUTCOMES:
Incidence of Nausea and vomiting will be described and treated accordingly. | Initiation of spinal anesthesia to 2 hrs after surgery
  0- no nausea no vomiting
  1. light nausea and no vomiting
  2. moderate nausea one or two vomiting episodes
  3. severe nausea, 3 or more vomiting episodes

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. BishnuPokharel, Dharān, Sunsari, Nepal

IPD SHARING:
Plan to Share IPD: No
I do not want to share IPD with other investigators

REFERENCES:
- [Background] Duncan CM, Hall Long K, Warner DO, Hebl JR. The economic implications of a multimodal analgesic regimen for patients undergoing major orthopedic surgery: a comparative study of direct costs. Reg Anesth Pain Med. 2009 Jul-Aug;34(4):301-7. doi: 10.1097/AAP.0b013e3181ac7f86. PMID 19574862
- [Background] Paul g. Barash clinical anesthesia 7th edition
- [Background] Panning B, Lehnhardt E, Mehler D. [Transient low frequency hearing loss following spinal anesthesia]. Anaesthesist. 1984 Dec;33(12):593-5. German. PMID 6528963
- [Background] Buvanendran A, McCarthy RJ, Kroin JS, Leong W, Perry P, Tuman KJ. Intrathecal magnesium prolongs fentanyl analgesia: a prospective, randomized, controlled trial. Anesth Analg. 2002 Sep;95(3):661-6, table of contents. doi: 10.1097/00000539-200209000-00031. PMID 12198056
- [Background] Carpenter RL, Caplan RA, Brown DL, Stephenson C, Wu R. Incidence and risk factors for side effects of spinal anesthesia. Anesthesiology. 1992 Jun;76(6):906-16. doi: 10.1097/00000542-199206000-00006. PMID 1599111
- [Background] Morikawa KI, Bonica JJ, Tucker GT, Murphy TM. Effect of acute hypovolaemia on lignocaine absorption and cardiovascular response following epidural block in dogs. Br J Anaesth. 1974 Sep;46(9):631-5. doi: 10.1093/bja/46.9.631. No abstract available. PMID 4621170
- [Background] Reiz S, Nath S, Ponten E, Friedman A, Backlund U, Olsson B, Rais O. Effects of thoracic epidural block and the beta-1-adrenoreceptor agonist prenalterol on the cardiovascular response to infrarenal aortic cross-clamping in man. Acta Anaesthesiol Scand. 1979 Oct;23(5):395-403. doi: 10.1111/j.1399-6576.1979.tb01466.x. PMID 43650
- [Background] Dobson PM, Caldicott LD, Gerrish SP, Cole JR, Channer KS. Changes in haemodynamic variables during transurethral resection of the prostate: comparison of general and spinal anaesthesia. Br J Anaesth. 1994 Mar;72(3):267-71. doi: 10.1093/bja/72.3.267. PMID 8130043
- [Background] Coe AJ, Revanas B. Is crystalloid preloading useful in spinal anaesthesia in the elderly? Anaesthesia. 1990 Mar;45(3):241-3. doi: 10.1111/j.1365-2044.1990.tb14696.x. PMID 2334037
- [Background] McCrae AF, Wildsmith JA. Prevention and treatment of hypotension during central neural block. Br J Anaesth. 1993 Jun;70(6):672-80. doi: 10.1093/bja/70.6.672. PMID 8329261
- [Background] Sigdel S. Prophylactic use of iv atropine for prevention of spinal anesthesia induced hypotension and bradycardia in elderly. A randomized controlled trial. J anesthesiol clin res.2015;4(1):5
- [Result] Stevens RD, Van Gessel E, Flory N, Fournier R, Gamulin Z. Lumbar plexus block reduces pain and blood loss associated with total hip arthroplasty. Anesthesiology. 2000 Jul;93(1):115-21. doi: 10.1097/00000542-200007000-00021. PMID 10861154